CLINICAL TRIAL: NCT00661427
Title: A Phase II Randomized Study of Cetuximab at Either 500 or 750 mg/m^2 Every Other Week for Recurrent or Metastatic Head and Neck Squamous Cell Cancer.
Brief Title: Cetuximab at Either 500 or 750 mg/m2 Every Other Week for Recurrent or Metastatic Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-039
Record Dates: First submitted 2008-01-07; First posted 2008-04-18 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Head and Neck; Squamous Cell Cancer
Keywords: Head and Neck cancer; Cetuximab
MeSH Terms: conditions — Neoplasms, Squamous Cell; Head and Neck Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab 500 mg/m^2 (Active Comparator): Cetuximab 500 mg/m^2 IV over 2 hours every other week
  Interventions: Biological: cetuximab
- Cetuximab 750 mg/m^2 (Active Comparator): Cetuximab 750 mg/m^2 IV over 3 hours every other week
  Interventions: Biological: cetuximab

INTERVENTIONS:
Biological: cetuximab — Cetuximab 500 mg/m^2 IV over 2 hours every other week
  Other Names: Erbitux
  Arms: Cetuximab 500 mg/m^2
Biological: cetuximab — Cetuximab 750 mg/m^2 IV over 3 hours every other week
  Other Names: Erbitux
  Arms: Cetuximab 750 mg/m^2

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, 2 doses of Cetuximab will have on head and neck cancer. The study is done because 250 mg/m2 given weekly does not work very well. Doses as high as 700 mg/m2 every other week appear to be no more toxic, so we will try to determine if 500 mg/m2 and 750 mg/m2 given every other week can work better. We do not know if it will help. We can use what we learn from this research study to help other people with the same disease.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent and HIPAA authorization
* histologically confirmed squamous cell cancer of the head and neck
* At least 21 days must have elapsed from the administration of prior chemotherapy for recurrent/metastatic disease.
* measurable disease as defined by RECIST
* ECOG PS ≤ 2
* Adequate hematologic function as defined by an ANC > or = to 1200/mm3 , and a platelet count ≥ 100,000 obtained within 14 days prior to enrollment.
* Adequate hepatic function as defined by t. bilirubin ≤ 1.5 mg/dl, transaminases & alk phos ≤ 5x ULN obtained within 14 days prior to enrollment.
* Adequate renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance >40 mL/minute.
* Women of childbearing potential must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study and have a negative pregnancy test within 7 days prior to registration. If a male and sexually active, the patient agrees to use effective contraception.
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.
* Patients with treated CNS metastases may be eligible if they have fully recovered from radiation therapy, surgery or steroids that were prescribed for CNS metastases.

Exclusion Criteria:

* Known, uncontrolled CNS metastases. CT/MRI of the brain is not required unless CNS metastases are suspected clinically.
* prior cetuximab therapy in the setting of recurrence or refractory disease
* Other active invasive malignancies, other than non-melanoma skin cancers or in situ cervical cancer.
* Concurrent treatment with other anti-cancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemo-embolization, or targeted therapy.
* Ongoing or active clinically serious infection > CTCAE Grade 2 requiring IV antibiotics, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia,(patients with stable rate-controlled atrial fibrillation may be eligible) or other medical condition that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study, or psychiatric illness/social situations that would limit compliance with study requirements.
* elective or planned major surgery to be performed during the course of the trial
* pregnant or lactating women
* employees of the investigator or study center w/ direct involvement in this study or other studies under the direction of the or study center, as well as family member of the employees
* More than two prior cytotoxic regimens for metastatic/recurrent disease.
* Known hypersensitivity reaction to mouse antibodies.
* Patients with nasopharyngeal cancer are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fury, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (17):
- United States (17):
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffit Cancer Center and Research Institute, Tampa, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York
  - Fox Chase Virtua Health Cancer Program, Philadelphia, Pennsylvania
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Abramson Cancer Center University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Huntsman Cancer Institue, Salt Lake City, Utah

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab Infusion at 500 mg/m^2: Cetuximab infusion at 500 mg/m^2 over 2 hours every other week.
- Cetuximab Infusion at 750 mg/m^2: Cetuximab infusion at 750 mg/m^2 over 3 hours every other week.
Period: Overall Study
Arm/Group | Cetuximab Infusion at 500 mg/m^2 | Cetuximab Infusion at 750 mg/m^2
Started | 35 | 26
Completed | 30 | 19
Not Completed | 5 | 7
Not completed — Adverse Event | 5 | 5
Not completed — Patient not treated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Cetuximab infusion at 500 mg/m2 over 2 hours every other week.
- Arm B: Cetuximab infusion at 750 mg/m2 over 3 hours every other week.
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 35 | 26 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 19 | 42
  >=65 years | 12 | 7 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Overall Objective Response
Description: Patients will be evaluated for response according to a modified version of the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines. Target lesions: Complete Response (CR): The disappearance of all target lesions. To be assigned a status of complete response, changes in tumor measurements must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. Partial Response (PR): At least a 30% decrease in the sum of the longest diameters of target lesions,taking as reference the baseline sum longest diameter. To be assigned a status of partial response, changes in tumor measurements must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify progressive disease. To be assigned a status of stable disease, taking as reference the smallest sum longest diam
Time Frame: Approximately every 8 weeks with imaging up to two years
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 30 | 19
participants
  Partial Response (PR) | 4 | 2
  Stable Disease (SD) | 12 | 5
  Progression of Disease (POD) | 14 | 12

2. Secondary Outcome: The Total Number of Participants That Were Effected by Adverse Events.
Description: Terminology Criteria Version 3.0 or study specific toxicity tables provided in the protocol define severity.
Time Frame: at least weekly
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 30 | 19
Participants | 28 | 18

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 18/30 | 7/19
Other Adverse Events (participants affected / at risk) | 28/30 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=30) | Arm B (N=19)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Allergic reaction (including drug fever) (General disorders) | 3 (3) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death not associated with CTCAE term- Death NOS (General disorders) | 2 (2) | 0 (0)
Death not associated with CTCAE term-Disease progression NOS (General disorders) | 4 (4) | 1 (1)
Dehydration (General disorders) | 2 (4) | 1 (1)
Dysphagia (Difficulty swallowing) (General disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ileus, GI (func obstruction of bowel) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Infection w/ Gr 3/4 neut, Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Nausea (General disorders) | 2 (2) | 0 (0)
Neuroendocrine: ADH secretion abnormal (Endocrine disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (5) | 0 (0)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Somnolence/depressd level of conscious (Psychiatric disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0)
Calcium, high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle weakness - Whole body/general (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=30) | Arm B (N=19)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anorexia (General disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dehydration (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (15) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Mood alteration - Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Mucositis (func/sympt)- Oral cavity (General disorders) | 2 (2) | 1 (1)
Muscle weakness - Whole body/general (General disorders) | 2 (2) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 14 (20) | 6 (6)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 11 (15) | 8 (9)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Trismus (General disorders) | 3 (3) | 1 (1)
Weight loss (General disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Taste alteration (dysgeusia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (fainting) (General disorders) | 0 (0) | 1 (1)
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (1)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Infection, other (Infections and infestations) | 0 (0) | 1 (1)
Inf norm ANC/gr1/2 neut (Infections and infestations) | 0 (0) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry mouth/salivary gland (xerostomia) (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
For safety data please see adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes